CLINICAL TRIAL: NCT06558929
Title: Evaluating the Effectiveness of Intervention Based on the Model of Occupational Harmony in Patients With Sleep Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOHar-CRSWD-001
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Circadian Rhythm Sleep-Wake Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occupational Intervention Group (Experimental): The intervention group will participate in a 6-week occupational therapy program, which includes 3 group treatment sessions, 1 individual treatment session, and daily occupational tasks.
  Interventions: Behavioral: Occupational Therapy; Other: Conventional Treatment

INTERVENTIONS:
Behavioral: Occupational Therapy — Participants will redesign their daily routine with support from occupational therapists and an online health management platform.
Other: Conventional Treatment — Participants will receive conventional treatment and education on sleep hygiene.

SUMMARY:
The goal of this clinical trial is to learn the effectiveness of an intervention based on the Model of Occupational Harmony (MOHar) in treating patients with sleep disorders. The main questions it aims to answer are:

* Does intervention based on the MOHar improve sleep quality in patients with sleep disorders?
* Does intervention based on the MOHar improve the quality of life in patients with sleep disorders?

Researchers will compare the intervention based on the MOHar to conventional treatment to see if the intervention works to treat sleep disorders.

Participants will:

* Participate in an occupational therapy program for 6 weeks (including group therapy, individual treatment, and daily occupational tasks)
* Complete questionnaires at 1, 3, and 6 months after the program for follow-up

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* self-reported difficulties with sleep quality
* active sleep disturbance as indicated by a PSQI > 5 or an ISI ≥ 8 at screening
* able to participate in research independently or with the assistance of a caregiver
* participate voluntarily in the study and sign an informed consent form

Exclusion Criteria:

* unable to cooperate with the study process due to cognitive, sensory, and motor dysfunction
* unable to skillfully use wearable monitoring devices or smartphones
* diagnosed with severe cardiac, liver, and kidney dysfunction and nervous system diseases
* have cardiac pacemakers
* being pregnant
* participating in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | 6 months
  Using the ISI to measure sleep quality
Pittsburgh Sleep Quality Index | 6 months
  Using the PSQI to measure sleep quality
36-Item Short Form Survey (SF-36) | 6 months
  Using the SF-36 to measure quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No